CLINICAL TRIAL: NCT01022697
Title: Randomized Control Study : Evaluation of the Benefits of Glucose Drinks During Childbirth
Brief Title: Evaluation of the Benefits of Glucose Drinks During Childbirth
Acronym: SOLISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007-A00585-48
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Childbirth

ARMS (2):
- A (Active Comparator): Glucose drink
  Interventions: Other: Glucose drink
- B (No Intervention): Fasting

INTERVENTIONS:
Other: Glucose drink — 200 mL each 3 hours up to 8 cm of dilatation
  Arms: A

SUMMARY:
Fear of full stomach when emergency general anaesthesia is required is the origin of fastening when giving birth. This behaviour does not warranty perfect security for the general anaesthesia. In addition, well being for women and new born is affected. Giving birth is finally compared to a sportive competition with high-energy needs. As Intravenous energy intake is not regulated by physiologic digestion, it can induce metabolic disorders for the mother that can be amplified for the foetus.

Oral glucose drinks could offer some benefits:

* gastric acidity would be decreased without significant increase in volumes.
* energy intake would further more active and more efficiency labour
* an increase in foetus well being

However, it has never been shown yet that such behaviour could offer those benefits. Also, it seems that there is not more vomiting, but most of the studies compared oral glucose intake to waterborne intake with the same volumes The expected efficacy is a reduction in labour duration and a reduction in percentage of extraction. Previous studies said that the lack of statistical power due to small number of subjects caused the absence of statistical significant relationship.

In addition, even though newborn have less acidosis, there is no clinical relationship proven.

The investigators propose a randomised multicentre study to assess efficacy of oral glucose drinks in comparison to traditional fastening when giving birth.

Main objective is to significantly reduce instrumental extraction rates. 5400 women will be included in the study in 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 yrs
* Entering for childbirth
* Informed written consent

Exclusion Criteria:

* more of 8 cm of dilatation
* Caesarean section planned
* natural delivery non-indicated
* pre-partum hemostasis troubles
* salicylic acid or anticoagulant treatment
* pre-eclampsia or HELLP syndrome
* diabetic neuropsy with troubles in gastric emptying
* IMC > 40 at the end of pregnancy
* understanding of the information
* under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4142 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Instrumental extraction rates | During childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse SIMONET, MD, Principal Investigator — University Hospital, Caen
Locations (9):
- France (9):
  - Hospital, Avranches, Avranches
  - Centre Hospitalier, Bayeux
  - Clinique du Parc, Caen
  - University Hospital, Caen, Caen
  - Centre Hospitalier du Rouvray, Elbeuf
  - University Hospital, Lille, Lille
  - Hospital, Mont Saint Aignan, Mont-Saint-Aignan
  - University Hospital, Rouen, Rouen
  - Centre Hospitalier Mémorial France Etats-Unis, Saint-Lô